CLINICAL TRIAL: NCT03503019
Title: Fructosamine as a Predictor of Surgical Outcomes in Total Joint Arthroplasty A Prospective Multi-center Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 18JPAR
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic
- Non-diabetic

SUMMARY:
A prospective multicenter study including all patients undergoing elective total hip (THA) or knee (TKA) arthroplasty (primary and revision). Patients will be screened for glycemic control using HbA1c levels, fructosamine levels, and blood glucose levels. Blood samples will be obtained at the preadmission testing (PAT) within 30 days of surgery. On postoperative day 1 (POD-1), morning glucose levels will be obtained for all patients as well. Patients will be followed up for 90 days postop.

Study aims

1. To examine the association between serum fructosamine levels and the risk for adverse outcomes (mainly PJI) following TJA among patients with and without diabetes.
2. To compare the utility of fructosamine levels to HbA1c in predicting adverse outcomes.
3. To determine the "best" threshold of fructosamine to determine adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

all patients undergoing elective total hip (THA) or knee (TKA) arthroplasty (primary and revision)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing elective total hip (THA) or knee (TKA) arthroplasty (primary and revision).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Joint Infection | within 90 days of surgery